CLINICAL TRIAL: NCT02645955
Title: Epidemiological Study of Hepatitis E Virus in Maintenance Hemodialysis Patients
Acronym: MHD HEV
Status: Completed | Type: Observational
Sponsor: Xiamen University (Other)
Responsible Party: Principal Investigator, Jun Zhang, vice-president of School of public health, Xiamen University
Other Study IDs: MHD-01
Record Dates: First submitted 2015-12-24; First posted 2016-01-05 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis E Virus Infection
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group, disease history: people who didn't have disease history of Maintenance Hemodialysis
- The MHD patient group, diseases history: Maintenance Hemodialysis Patients

SUMMARY:
Primary Purpose:

1. Evaluate the prevalence and incidence of HEV infection in MHD patients.
2. Compare differences of the prevalence and incidence between the MHD patients and the control. .

Secondary purpose:

Analyze risk factors of HEV infection.

DETAILED DESCRIPTION:
This is an Epidemiological study manufactured by Xiamen University. The primary purpose of this study is to evaluate the prevalence and incidence of HEV infection in MHD patients and to compare differences between the MHD patients and the control. The secondary purpose of this study is to analyze risk factors of the infection of HEV. There are two phases in this study. The first phase is a cross-sectional study. Approximately 200 MHD patients will be enrolled in MHD patient group, followed by control group's enrollment according to the age and gender of the MHD patient group. Blood samples and questionnaire were got at this time. Secondly, 100 enrolled volunteers in each group who is negative for HEV-IgM、HEV-IgG、HEV RNA will be introduced into the cohort study. The MHD patient group will been taken blood samples at an interval of 3 month until the 12th month after the first phase, however, the control group only need one blood sample at 12th month.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis patients and healthy people as control
* Can understand the study progress, willing to sign the informed consent and participate the study

Exclusion Criteria:

* Has received HEV vaccines

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 200 each for the MHD patient group and the control group
Sampling Method: Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
prevalence of HEV infection | up to 1 year after enrollment
  number and rate of participants with abnormal laboratory values in the MHD patients and the control;
new-infection rate of HEV infection | up to 1 year after enrollment
  number and rate of the participants who's baseline laboratory value is normal and change to abnormal during the follow-up in the MHD patients and the control

SECONDARY OUTCOMES:
risk factors of HEV infection | up to 1 year after enrollment
  the odd ratio(OR) and 95%CI of the factors such as age gender for HEV infection in the MHD patients and the control

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Niu, M.Sc., Principal Investigator — Zhongshan Hospital Xiamen University